CLINICAL TRIAL: NCT05641844
Title: A Prospective, Multi-Center, Double Blind, Randomized Controlled Study, Evaluating the Safety and Efficacy of RD2 Ver.02, For the Management of Anal Fistulas
Brief Title: A Double Blind, Randomized Controlled Study, Evaluating the Safety and Efficacy of RD2 Ver.02 For the Management of Anal Fistulas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RedDress Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RD014
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment arm (Other): Subjects will undergo debridement of the fistula tract and suturing of internal opening, followed by a. water leak test. RD2 Ver.02 will be applied to the fistula tract in the operating room.
  Interventions: Device: RD2 Ver.02; Other: Saline
- Control arm (Other): Subjects will undergo debridement of the fistula tract and suturing of internal opening, followed by a. water leak test. Saline will be applied to the fistula tract in the operating room.
  Interventions: Other: Saline

INTERVENTIONS:
Device: RD2 Ver.02 — Debridement and suturing of the internal opening of the anal fistula and RD2 Ver.02 coagulating blood application into the fistula tract with a semi flexible cannula.
  Arms: Treatment arm
Other: Saline — Debridement and suturing of the internal opening of the anal fistula and Saline administration into the fistula tract with a semi flexible cannula.

SUMMARY:
The goal of this clinical trial is to assesses the safety of autologous RD2 Ver.02 as compared to a control for managing transsphincteric and intersphinsteric anal fistulas.

The main questions it aims to answer are:

Assess the safety and efficacy of RD2 Ver.02 in anal fistula application, compared to control.

Complication rate by 6 months of anal fistula treatment with RD2 Ver.02 compared to control.

Recurrence of anal fistula at 12 months post-treatment Incidence of perirectal infection by 6 months in anal fistulas treated with RD2 Ver.02 compared to control.

Patients will be randomized in to 2 arms. For all patients, blood will be drawn to ensure the blinding of the patients, the fistula will be evaluated and debrided, and then the internal fistula opening will be suture-closed, and a water leak test will be performed to ensure sealing. Following the water leak test, In the treatment arm, the patient's own coagulating blood will be applied into the entire fistula tract, allowing it to clot and serve as a provisional matrix inside the fistula tract. In the control arm, the blood sample will be discarded and saline will be applied to the fistula tract.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years of age
* Subject has a transsphincteric or long intersphincteric anal fistula (>1.5 cm), with a seton in place for a minimum of 1 month, deemed eligible for primary or repeat fistula repair by anorectal advancement flap or LIFT: Anterior, posterior or lateral fistula, first or recurrent, at any position circumferentially, with one external opening and one internal opening.
* Subjects is unable or unwilling to receive invasive surgical procedures, anorectal advancement flap or LIFT procedure, and is opting for minimally invasive technique of anal fistula management (i.e., fistula tract debridement and suturing of internal opening).
* 2.1.4 Prior to enrollment, during the preceding 3 months from Treatment Visit, subject must undergo a pelvic MRI to evaluate eligibility criteria unable to be assessed clinically.
* Female subjects who are capable of conceiving and all males capable of insemination must use an acceptable form of contraception in order to participate in the study and for 6 months following study procedure (acceptable forms of contraception include condoms for males and contraceptive pills or IUDs for women)

Exclusion Criteria:

* Subject who has a life expectancy of less than 24 months.
* Subjects who are cognitively impaired and have a healthcare proxy or those who are cognitively impaired and clearly do not understand the contents of the informed consent form.
* Cannot withdraw blood in the required amount (up to 15 mL).
* Women who are pregnant or currently breast feeding.
* Subject is currently receiving (i.e., within the past 30 days) or scheduled to receive systemic steroids (more than 10mg per day).
* Multiple fistula tracts, as confirmed on pelvic MRI
* Short fistula tract that in the surgeon's opinion are amenable to fistulotomy
* Active infection including perianal infection, and/or any active systemic or local infection.
* Presence of a perirectal abscess on pelvic MRI
* Presence of dominant luminal active Crohn's disease, validated by recent colonoscopy from preceding 12 months, requiring immediate therapy
* Rectal and/or anal stenosis and / or active proctitis, if this means a limitation for any surgical procedure.
* Known allergies or hypersensitivity to any of the following: antibiotics including but not limited to penicillin, streptomycin, gentamicin, aminoglycosides; Human Serum Albumin (HSA); Dulbecco Modified Eagle's Medium (DMEM); materials of bovine origin; local anaesthetics or gadolinium (MRI contrast); Known hypersensitivity to reagents and components of RD2 Ver.02 including calcium gluconate, Kaolin or citrate and ethylene oxide.
* Contraindication to MRI scan, (e.g., due to the presence of pacemakers, hip replacements, or severe claustrophobia).
* Known coagulation problems, abnormal thrombocytes level or if heparin is given intravenously. Subjects who are taking Coumadin, Aspirin, Plavix (Clopidogrel), Eliquis or Pradaxa will not be excluded.
* Patients with increased risk for the surgical procedure or major alteration of any of the following laboratory tests:

  1. Serum Creatinine levels >1.5 times the upper limit of normality (ULN)
  2. Total bilirubin >1.5 times the ULN (unless predominantly non conjugated due to documented history of Gilbert's syndrome)
  3. AST/ ALT >3.0 times the ULN
  4. Hemoglobin <10.0 g/dL
  5. Platelets <150.0 x109/L
  6. Albuminemia <3.0 g/dL.
* Patients who do not wish to or cannot comply with study procedures.
* Patients currently receiving or having received within 12 months prior to enrolment into this clinical study, any investigational drug.
* Subjects who need surgery in the perianal region for reasons other than fistulas at the time of inclusion in the study, or for whom such surgery is foreseen in this region in the 24 weeks after treatment administration.
* Contraindication to the anesthetic procedure.
* Subject with a diagnosis of Ulcerative Colitis
* Subject with malignancy, undergoing active treatment
* Rectovaginal fistula
* History of pelvic radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Combined healing rate at 6 months of anal fistulas treated with RD2 Ver.02 compared to control | 6 months after anal fistula treatment per subject
  Fistula healing will be assessed by both a blinded clinical assessor and confirmation by MRI. Healing clinical assessment is defined as the absence of any anal symptom, with no discharge from the fistula and a closed external opening. Results will be confirmed by central blinded MRI assessment.

SECONDARY OUTCOMES:
Clinical recurrence of anal fistula at 12 months post-treatment in subjects with clinically healed fistula at 6 months, treated with RD2 Ver. 02 compared to control, to evaluate the long-term efficacy of RD2 Ver.02 Application. | 12 months
  Assessed by the blinded clinical assessor for fistula recurrence 12 months post procedure
Incidence of perirectal infection by 6 months in anal fistulas treated with RD2 Ver.02 compared to control. | 6 months
  Infection assessment of the anal fistula

OTHER OUTCOMES:
Incidence of device-related adverse events in patients treated with RD2 Ver.02 | 12 months
  Overall incidence and severity of Adverse Events (AEs) in RD2 Ver.02 treatment group
Incidence of adverse events compared between RD2 Ver.02 and control arms | 12 months
  Comparison of the AEs between RD2 Ver.02 and control treatment groups

CONTACTS AND LOCATIONS:
Locations (10):
- United States (9):
  - Karen Zaghiyan, M.D, Los Angeles, California
  - Cleveland Clinic, Weston, Florida
  - University of Chicago, Chicago, Illinois
  - Franciscan Health, Indianapolis, Indiana
  - UMASS, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Lenox Hill Hospital, New York, New York
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Brown surgical associates, Providence, Rhode Island
- Sheba Medical Center, Ramat Gan, Israel